CLINICAL TRIAL: NCT00786240
Title: A Phase 1, Open-Label, Randomized, Single-Dose, 2-Way Crossover Study To Determine Bioequivalence Of 4 Mg Fesoterodine SR Tablet Between Formulation D And Formulation E(1) In Healthy Subjects.
Brief Title: Phase1, Single Dose, Crossover Study to Determine Bioequivalence
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: A0221063
Record Dates: First submitted 2008-11-05; First posted 2008-11-06 (Estimated); Last update posted 2010-09-09 (Estimated); Status verified 2010-09

CONDITIONS: Healthy
Keywords: Bioequivalence; Therapeutic Equivalency
MeSH Terms: interventions — fesoterodine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental)
  Interventions: Drug: Fesoterodine
- B (Experimental)
  Interventions: Drug: Fesoterodine

INTERVENTIONS:
Drug: Fesoterodine — Single dose of 4 mg tablet in formulation D under fasted conditions (Reference)
  Arms: A
Drug: Fesoterodine — Single dose of 4 mg tablet in formulation E(1) under fasted conditions (Test)
  Arms: B

SUMMARY:
The objective of this study is to demonstrate bioequivalence of 4 mg tablet of formulation D and formulation E(1).

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female Chinese or Japanese subjects

Exclusion Criteria:

* Evidence or history of clinically significant findings at screening

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 37 (Actual)
Dates: Start 2009-01; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
AUCt and Cmax of 5-HMT after single oral administration of 4 mg fesoterodine SR tablets in formulation D under fasted conditions | Day 1 and 2
AUCt and Cmax of 5-HMT after single oral administration of 4 mg fesoterodine SR tablets in formulation E(1) under fasted conditions | Day 1 and 2

SECONDARY OUTCOMES:
Tmax, AUClast, AUCinf, kel, t½ and MRT after single oral administration of 4 mg fesoterodine SR tablets in formulation D under fasted conditions | Day 1 and 2
Tmax, AUClast, AUCinf, kel, t½ and MRT after single oral administration of 4 mg fesoterodine SR tablets in formulation E(1) under fasted conditions | Day 1 and 2

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Singapore, Singapore, Singapore

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A0221063&StudyName=Phase1%2C%20single%20dose%2C%20crossover%20study%20to%20determine%20bioequivalence